CLINICAL TRIAL: NCT05863585
Title: An Open-Label Study to Evaluate the Safety and Immunogenicity of 2 Doses of 100µg BG505 SOSIP.664 gp140 Vaccine, Adjuvanted, Given to a Population of Adults in Good General Health Who Have Received 3 Doses of 300µg BG505 SOSIP.GT1.1 gp140 Vaccine, Adjuvanted
Brief Title: A Clinical Trial to Evaluate the Safety and Immunogenicity of a Prophylactic HIV Vaccine Candidate
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: International AIDS Vaccine Initiative (Network)
Collaborators: Access to Advanced Health Institute (AAHI) (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IAVI C107
Record Dates: First submitted 2023-04-07; First posted 2023-05-18 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Hiv
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — aluminum sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BG505 SOSIP.664 gp140 Vaccine, Adjuvanted (3M-052 AF plus alum) (Experimental): BG505 SOSIP.664 gp140 Vaccine, Adjuvanted (3M-052 AF plus alum) Dosage
  Interventions: Drug: BG505 SOSIP.664 gp140 Vaccine, Adjuvanted (3M-052 AF plus alum)

INTERVENTIONS:
Drug: BG505 SOSIP.664 gp140 Vaccine, Adjuvanted (3M-052 AF plus alum) — 100µg

SUMMARY:
An Open-Label Study to Evaluate the Safety and Immunogenicity of 2 Doses of 100µg BG505 SOSIP.664 gp140 Vaccine, Adjuvanted, given to a Population of Adults in Good General Health Who have Received 3 doses of 300µg BG505 SOSIP.GT1.1 gp140 Vaccine, Adjuvanted

DETAILED DESCRIPTION:
This is an open-label study to evaluate the safety and immunogenicity of 2 doses of 100µg of BG505 SOSIP.664 gp140 Vaccine, Adjuvanted, given to HIV-1 uninfected adults in good general health who have received 3 doses of 300µg BG505 SOSIP.GT1.1 gp140 Vaccine, Adjuvanted, as part of Protocol IAVI C101 (NCT04224701).

Up to 14 participants, who had enrolled in and completed the phase 1 Protocol IAVI C101 "A Clinical Trial to Evaluate the Safety and Immunogenicity of Recombinant HIV-1 Envelope Protein BG505 SOSIP.GT1.1 gp140 Vaccine, Adjuvanted in Healthy, HIV-uninfected Adults (NCT04224701) and who received 3 doses of 300µg of BG505 SOSIP.GT1.1 gp140 Vaccine, Adjuvanted, will be recruited into the study. Protocol IAVI C101 evaluated the capacity of GT1.1 to prime desirable on-target responses against the CD4 binding site (CD4bs) of the HIV virion, including but not limited to VRC01 class responses, as well as against V2-apex.

This study, Protocol IAVI C107, will examine if maturation of anti-HIV antibody response occurs following boost immunizations with BG505 SOSIP.664 gp140 Vaccine, Adjuvanted. It is expected that this study will provide insight into if and how BG505 SOSIP.664 immunization can expand and mature desirable on-target CD4bs and V1V2-apex responses.

ELIGIBILITY:
Inclusion:

* Healthy adults as assessed by a medical history, physical exam, and laboratory tests
* Received 3 doses of 300µg of BG505 SOSIP.GT1.1 gp140 Vaccine, Adjuvanted
* Willing to comply with the requirements of the protocol and be available for follow-up for the planned duration of the study
* In the opinion of the Principal Investigator (PI) or designee and based on Assessment of Understanding (AOU) results, has understood the information provided and potential impact and/or risks linked to vaccine administration and participation in the trial; written informed consent will be obtained from the participant before any study-related procedures are performed
* Willing to undergo HIV testing, risk reduction counseling and receive HIV-test results
* All participants born female who are engaging in sexual activity that could lead to pregnancy must commit to use an effective method of contraception starting 2 weeks before the first vaccine administration and for 4 months following the last vaccine administration. Effective contraception includes:
* Condoms (male or female) with or without spermicide
* Diaphragm or cervical cap with spermicide
* Intrauterine device
* Hormonal contraception, including contraceptive implant or injectable
* Oral contraception
* Successful vasectomy in the male partner

Considered successful if a woman reports that a male partner has:

1. documentation of azoospermia by microscopy (1 year ago) or
2. a vasectomy more than 2 years ago with no resultant pregnancy despite sexual activity post vasectomy • Not of reproductive potential Such as having undergone hysterectomy, bilateral oophorectomy, or tubal ligation, postmenopausal (≥45 years of age with amenorrhea for at least 2 years, or any age with amenorrhea for at least 6 months and a serum follicle stimulating hormone (FSH) level > 40 IU/L), surgically sterile Note: More restrictive measures may be required by the study sites. 7. All participants born female who are not heterosexually active at screening must agree to utilize an effective method of contraception if they become heterosexually active as outlined above 8. All participants born female must be willing to undergo urine pregnancy tests at time points indicated in the Schedule of Assessments (SOA) (Appendix A) 9. Willing to forgo donations of blood, or any other tissues during the study and, for those who test HIV-positive due to vaccine-induced antibodies, until the anti-HIV-antibody titers become undetectable

Exclusion Criteria

* Confirmed HIV-1 or HIV-2 infection
* Any clinically relevant abnormality on history or examination, including history of immunodeficiency or autoimmune disease; use of systemic corticosteroids (the use of topical or inhaled steroids is permitted), immunosuppressive, anticancer, anti-tuberculosis or other medications considered significant by the Investigator within the previous 6 months.

Note: The following exceptions are permitted and will not exclude study participation: use of corticosteroid nasal spray for rhinitis, topical corticosteroids for an acute uncomplicated dermatitis; or a short course (duration of 10 days or less, or a single injection) of corticosteroid for a non-chronic condition (based on Investigator clinical judgment) at least 2 weeks prior to enrollment in this study.

* Any clinically significant acute or chronic medical condition that is considered progressive or in the opinion of the Investigator makes the participant unsuitable for participation in the study
* Reported behavior that put the participant at risk for HIV infection within 6 months prior to vaccine administration, as defined by:
* Unprotected sexual intercourse with a known HIV-infected person, a partner known to be at high risk for HIV infection or a casual partner (ie, no continuing established relationship)
* Engaged in sex work
* Frequent excessive daily alcohol use or frequent binge drinking, or any other use of illicit drugs
* History of newly acquired syphilis, gonorrhea, non-gonococcal urethritis, HSV-2, chlamydia, pelvic inflammatory disease, trichomonas, mucopurulent cervicitis, epididymitis, proctitis, lymphogranuloma venereum, chancroid, or hepatitis B or hepatitis C
* Three or more sexual partners
* If female, pregnant, lactating, or planning a pregnancy during the period of enrollment until 4 months after the last vaccine administration
* Bleeding disorder that was diagnosed by a physician (eg, clotting factor deficiency, coagulopathy or platelet disorder that requires special precautions) Note: A participant who states that he/she has easy bruising or bleeding, but does not have a formal diagnosis and has IM injections and blood draws without any adverse experience is eligible
* Infectious disease diagnosis: chronic hepatitis B infection (HbsAg-positive), current hepatitis C infection (HCV Ab positive and HCV ribonucleic acid (RNA) positive or interferon-alfa treatment for hepatitis C infection in the past year or interferon-alfa-free treatment for hepatitis C infection completed in the past 6 months), or active syphilis (screening and confirmatory tests)
* History of splenectomy
* Any of the following abnormal laboratory parameters listed below:

Hematology

* Hemoglobin - <10.5 g/dl or <6.5 mmol/L in females; <11.0 g/dl or <6.8 mmol/L in males
* Absolute Neutrophil Count (ANC) - ≤1,000/mm3 or < 1.0 x 109 cells/L
* Absolute Lymphocyte Count (ALC) - ≤650/mm3 or < 0.65 x 109 cells/L
* Platelets - <125,000 cells/mm3 or <125 x 109 cells/L Chemistry
* Creatinine - >1.1 x upper limit of normal (ULN)
* AST - >1.25 x ULN
* ALT - >1.25 x ULN Urinalysis

Clinically significant abnormal dipstick confirmed by microscopy:

* Protein = 1+ or more
* Blood = 2+ or more (not due to menses)
* Receipt of live attenuated vaccine within the previous 30 days or planned receipt within 30 days after vaccine administration; or receipt of other vaccine within the previous 14 days or planned receipt within 14 days after vaccine administration. (Exception is live attenuated influenza vaccine within 14 days.)
* Receipt of blood transfusion or blood-derived products within the previous 3 months
* Participation in another clinical trial of a vaccine currently, within the previous 3 months or expected participation during this study (with the exception of Protocol IAVI C101); concurrent participation in an observational trial not requiring blood or tissue sample collection is not an exclusion
* Prior receipt of any investigational HIV vaccine candidate or HIV monoclonal antibody other than BG505 SOSIP.GT1.1 gp140 Vaccine, Adjuvanted
* History of significant local or systemic reactogenicity to vaccines (eg, anaphylaxis, respiratory difficulties, angioedema, injection site necrosis or ulceration)
* Psychiatric condition that compromises safety of the participant and precludes compliance with the protocol. Specifically excluded are persons with psychoses within the past 3 years, ongoing risk for suicide, or history of suicide attempt or gesture within the past 3 years
* Seizure disorder: A participant who has had a seizure in the last 3 years is excluded. (Not excluded: a participant with a history of seizures who has neither required medications nor had a seizure for 3 years)
* History of malignancy in the past 5 years (prior to screening) or ongoing malignancy (a history of completely excised malignancy, which is considered cured, is not an exclusion)
* Active, serious infections requiring antibiotic, antiviral, or antifungal therapy within 30 days prior to enrollment
* Body mass index (BMI) ≥35
* Body weight <110 pounds (50 kg)
* Prior daily use of NSAID/aspirin that cannot be held for 5 days prior to the leukapheresis procedure (if required by the study site)
* If, in the opinion of the PI, it is not in the best interest of the participant to participate in the trial

Ages: 18 Years to 51 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
To evaluate safety and tolerability of BG505 SOSIP.664 gp140 Vaccine, Adjuvanted (3M-052 AF plus alum) | 7 days
  Proportion of participants with Grade 2 or greater reactogenicity (ie, solicited AEs) from Day 0 through Day 7 after each vaccine administration
To evaluate safety and tolerability of BG505 SOSIP.664 gp140 Vaccine, Adjuvanted (3M-052 AF plus alum) | 28 days
  Proportion of participants with vaccine-related unsolicited AEs, including safety laboratory (biochemical, hematological) parameters, from the day of each vaccine administration up to 28 days post each vaccine administration
To evaluate safety and tolerability of BG505 SOSIP.664 gp140 Vaccine, Adjuvanted (3M-052 AF plus alum) | 28 days
  Proportion of participants with Grade 2 or greater unsolicited AEs, including safety laboratory (biochemical, hematological) parameters, from the day of each vaccine administration up to 28 days post each vaccine administration
To evaluate safety and tolerability of BG505 SOSIP.664 gp140 Vaccine, Adjuvanted (3M-052 AF plus alum) | 1 year
  Proportion of participants with vaccine-related SAEs throughout the study period
To evaluate safety and tolerability of BG505 SOSIP.664 gp140 Vaccine, Adjuvanted (3M-052 AF plus alum) | 1 year
  Proportion of participants in each group with potential immune-mediated diseases (pIMDs) from the day of first vaccine administration throughout the study period

SECONDARY OUTCOMES:
To determine the immunogenicity of BG505 SOSIP.664 gp140 Vaccine, Adjuvanted (3M-052 AF plus alum) | 1 year
  Frequency and magnitude of binding antibody responses to 2 doses of 100µg of BG505 SOSIP.664 gp140 Vaccine, Adjuvanted, given to adults in good general health who have received 3 doses of 300ug of BG505 SOSIP.GT1.1 gp140 Vaccine, Adjuvanted